CLINICAL TRIAL: NCT02137798
Title: Atrial Fibrillation Ablation Facilitated by Fluoroscopy Image Integrated 3-dimentional Electroanatomical Mapping System
Brief Title: Reduction of Fluoroscopy Exposure During Atrial Fibrillation Ablation
Acronym: AF-FII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Christopher Piorkowski, M.D., Technische Universität Dresden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EK474122013; CARTOUNIVU (Other Grant/Funding Number: Biosense Webster)
Record Dates: First submitted 2014-05-02; First posted 2014-05-14 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Atrial Fibrillation
Keywords: fluoroscopy exposure; paroxysmal atrial fibrillation Ablation; fluoroscopy; Atrial Fibrillation Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CARTOUNIVU (Experimental): Radiofrequency catheter ablation of atrial fibrillation will be performed using fluoroscopy image integrated 3-dimentional electroanatomical mapping system
  Interventions: Device: Radio-frequency catheter ablation
- CARTO3 (Active Comparator): Radiofrequency catheter ablation of atrial fibrillation will be performed using 3-dimentional electroanatomical mapping system without fluoroscopy image integration technique
  Interventions: Device: Radio-frequency catheter ablation

INTERVENTIONS:
Device: Radio-frequency catheter ablation — Radio-frequency atrial fibrillation catheter ablation includes circumferential PV isolation and voltage-map guided substrate modification, which means low voltage zone (amplitude < o.5 mV) will also be ablated.

SUMMARY:
To evaluate reduction of fluoroscopy time/dosis and safety of atrial fibrillation ablation in patients with paroxysmal atrial fibrillation using fluoroscopy image integrated 3-dimentional electroanatomical mapping system, comparing to using 3-dimentional electroanatomical mapping system without fluoroscopy image integration

DETAILED DESCRIPTION:
The novel fluoroscopic image integrated 3-dimentional electroanatomical mapping system is designed for minimizing the exposure to X-ray for physician, staff and patients. This randomized single-center study is to evaluate the reduction on fluoroscopy levels (time and dosis) in catheter interventional treatment of symptomatic, antiarrhythmic refractory paroxysmal atrial fibrillation using fluoroscopic image integrated 3-dimentional electroanatomical mapping system, comparing with using 3-dimentional electroanatomical mapping system without fluoroscopic image integration. Patients with documented paroxysmal atrial fibrillation, who are going to receive a catheter interventional treatment to atrial fibrillation, will be randomized (1:1) into two groups after signing an informed consent. Group 1 (CARTOUNIVU): using fluoroscopic image integrated 3-dimentional electroanatomical mapping system. Group 2 (CARTO3): using 3-dimentional electroanatomical mapping system without fluoroscopic image integration.

The ablation strategies in both study groups are the same, including circumferential isolation of ipsilateral pulmonary veins (PV) and voltage map guided substrate modification. According to the randomization, the ablation procedure will be performed with or without fluoroscopic image integration.

The primary endpoint of this study is the evaluation of reduction on fluoroscopy levels (fluoroscopy time and dosis) during atrial fibrillation ablation procedure. Secondary endpoints include complete isolation of the pulmonary veins, completely bidirectional block of linear ablation lines, total procedure time, ablation-related complications.

ELIGIBILITY:
Inclusion Criteria:

* documented atrial fibrillation in the 12-lead ECG or Holter ECG
* Paroxysmal symptomatic atrial fibrillation
* Ineffectiveness of antiarrhythmic medication ( at least 1 medication )
* Age 18-75 years
* left atrial diameter <60 mm ( Transesophageal Echocardiography, parasternal )
* A signed consent form

Exclusion Criteria:

* Reversible etiology of atrial fibrillation
* Pregnancy
* Women of childbearing potential without a negative pregnancy test within 48 hours prior to the ablation procedure
* Intracardiac thrombus
* Contraindication to anticoagulation
* Thromboembolic event in the last 6 months
* Previous left atrial ablation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Fluoroscopy time for each step of atrial fibrillation ablation procedure | 1 day ( at the end of each step of atrial fibrillation ablation procedure)
  Fluoroscopy time will be recorded at the end of each step of atrial fibrillation ablation, including femoral vein puncture, placement of catheters, transseptal puncture, system registration, reconstruction of left atrium, PV-Angiography, acquirement of voltage map, PV-isolation, confirmation of complete PV isolation and linear ablations.
Fluoroscopy doses for each step of atrial fibrillation ablation procedure | 1 day ( at the end of each step of atrial fibrillation ablation procedure)
  Fluoroscopy doses will be recorded at the end of each step of atrial fibrillation ablation, including femoral vein puncture, placement of catheters, transseptal puncture, system registration, reconstruction of left atrium, PV-Angiography, acquirement of voltage map, PV-isolation, confirmation of complete PV isolation and linear ablations.

SECONDARY OUTCOMES:
Number of patients with adverse events as a measure of safety | All patients will be followed for the duration of hospital stay for acute complications, an expected average of 3 days.
  Perforation, tamponed, phrenic nerve injury and oesophagus injury (patients will be screened for oesophagus injury for a month after atrial fibrillation ablation), etc.
Number of patients with a failure of reaching endpoints of procedure as a measure of efficacy | 1 day ( at the end of each step of atrial fibrillation ablation procedure)
  number of pulmonary veins/linear ablation lines has not been completely isolated/blocked at the end of the AF ablation
Total time of atrial fibrillation ablation procedure as a measure of efficacy | up to 24 hours
  procedure time (minute)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Piorkowski, M.D., Principal Investigator — Department of Electrophysiology, University of Dresden - Heart Center
Locations (1):
- Department of Electrophysiology, University of Dresden - Heart Center, Dresden, Saxony, Germany